CLINICAL TRIAL: NCT02036476
Title: Cabozantinib in Recurrent/Metastatic Merkel Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Principal Investigator, Robert Haddad, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-490
Record Dates: First submitted 2013-12-19; First posted 2014-01-15 (Estimated); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Merkel Cell Carcinoma; Skin Cancer
Keywords: Merkel Cell Carcinoma; Skin Cancer
MeSH Terms: conditions — Carcinoma, Merkel Cell; Skin Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabozantinib (Experimental): Cabozantinib 60 mg given orally daily for 28 days (4 weeks) each cycle. Participants were treated until disease progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — oral administration
  Other Names: XL184; Cometriq

SUMMARY:
This is an open-label, non-randomized, phase 2 study to assess the feasibility of using cabozantinib in recurrent/metastatic Merkel Cell Carcinoma patients that progressed after platinum-based therapy.

DETAILED DESCRIPTION:
Cabozantinib (XL184) is an inhibitor of multiple receptor tyrosine kinases and was approved by the U.S. Food and Drug Administration (FDA) on 29 November 2012 for the treatment of patients with progressive, metastatic medullary thyroid cancer. It is commercially available as COMETRIQ™ in the United States.

During the Pre Treatment Period, participants are consented and qualified (screened) for the study. Treatment will be administered on an outpatient basis.

Each treatment cycle lasts 28 days, during which time the participant will be taking the study drug, cabozantinib, once daily. The participant will be given a study drug-dosing diary for each treatment cycle. The diary will also include special instructions for taking the study drug.

- Participants will be followed for 8 weeks after removal from study or until death, whichever occurs first. Participants removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed Merkel Cell Carcinoma that is metastatic or unresectable and for which standard curative measures do not exist or are no longer effective
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥10 mm with spiral CT scan (see section 10 for the evaluation of measureable disease). Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented
* Must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin or another organoplatinum compound. Patients are also eligible if they received curative intent platinum-based therapy and progressed within a year of therapy
* No prior MET inhibitor is allowed
* At least 2 weeks since prior chemotherapy or radiation therapy. At least 3 weeks since prior biologics or investigational agents
* Recovery from effects of recent treatment to baseline or CTCAE ≤ grade 1 toxicity from all prior therapies except alopecia and other non-clinically significant AEs
* Participants must be ≥18 years of age
* ECOG performance status ≤1
* Participants must have normal organ and marrow function
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation
* Ability to understand and the willingness to sign a written informed consent document
* Collection of archival tissue specimens for confirmation of Merkel Cell Carcinoma

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier
* Participants may not be receiving any biologics or investigational agents within 3 weeks
* The subject has active brain metastases or epidural disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cabozantinib
* Has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test ≥ 1.3 the institutional ULN within 7 days before the first dose of study treatment, unless PT/PTT prolongation known to be secondary to conditions not associated with increased bleeding risk (as on antiphospholipid antibody syndrome)
* Requires concomitant treatment, in therapeutic doses, with anticoagulants
* Active bleeding or pathologic conditions that carry high risk of bleeding
* Have experienced clinically significant gastrointestinal bleeding within 6 months before first dose of study treatment
* Requires chronic concomitant treatment of strong CYP3A4 inducers
* Is unable or unwilling to swallow tablets
* Has a corrected QT interval calculated by the Fridericia formula (QTcF)>500 ms within 28 days before initiation of cabozantinib
* Has evidence of tumor invading the GI tract or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* Has radiographic evidence of cavitating pulmonary lesion(s)
* Has uncontrolled, significant intercurrent or recent illness
* Other disorders associated with a high risk of fistula formation including PEG tube placement within 3 months before the first dose of study therapy
* History of major surgery within 3 months or minor surgery within 1 month of the first dose of cabozantinib
* Pregnant women
* Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy
* HIV-positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Haddad, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data. Cumulative results will be posted here and published.

REFERENCES:
- [Result] Rabinowits G, Lezcano C, Catalano PJ, McHugh P, Becker H, Reilly MM, Huang J, Tyagi A, Thakuria M, Bresler SC, Sholl LM, Shapiro GI, Haddad R, DeCaprio JA. Cabozantinib in Patients with Advanced Merkel Cell Carcinoma. Oncologist. 2018 Jul;23(7):814-821. doi: 10.1634/theoncologist.2017-0552. Epub 2018 Feb 14. PMID 29445030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from February 2014 to March 2016.
Groups:
- Cabozantinib: Cabozantinib 60 mg Oral Daily 28 days (4 weeks)
Period: Overall Study
Arm/Group | Cabozantinib
Started | 8
Completed | 0
Not Completed | 8
Not completed — Withdrawal by Subject | 2
Not completed — Progressive Disease | 4
Not completed — Unacceptable Toxicity | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 2
  White | 6

OUTCOME MEASURES:

1. Primary Outcome: 3-Month Disease Control Rate (DCR)
Description: 3-month DCR is the percentage of participants achieving complete response (CR), partial response (PR) or stable disease (SD) during first 3 months of treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PD is at least a 20% increase in sum LD of target lesions (smallest sum LD reference), new lesions, and/or unequivocal progression of existing non-target lesions. Stable disease (SD) is defined as any condition not meeting the above criteria and lasting at least 3 months from baseline.
Time Frame: Disease was assessed on day 1 of weeks 3, 5, 7, 9, 11, 13 then every 4 weeks on treatment. Relative to this endpoint was observation up to 3 months on treatment. Length of longest follow up was 83 days.
Population: The analysis population is all enrolled participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 8
percentage of participants | 12.5 [0.64 to 47.07]

2. Secondary Outcome: 3-month Progression-free Survival (PFS)
Description: 3-month PFS is a probability based on the Kaplan-Meier (KM) method. PFS is defined as the duration of time from registration to documented disease progression (PD) or death, or censored at date of last disease assessment. Per RECIST v1.1: PD is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Assessed every 2 weeks (w) from cycles 3-13 and then every 4w, day 30-37 post-treatment end and up to 8w in long-term follow-up. Length of longest follow up for the KM estimate was 126 days. Relative to this endpoint was 3-month probability.
Population: The analysis population is all enrolled participants.
Measure: Number (90% Confidence Interval); unit: probability
Arm/Group | Cabozantinib
Number analyzed (Participants) | 8
probability | 0.19 [0.046 to 0.81]

3. Secondary Outcome: 3-Month Overall Survival (OS) Rate
Description: 3-month OS rate is the percentage of patients alive at 3 months from registration.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 8
percentage of participants | 100 [65 to 100]

4. Secondary Outcome: Grade 3-5 Treatment-Related Adverse Event (AE) Rate
Description: All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Rate is the percentage of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation.
Time Frame: Up to 126 days
Population: The analysis population is all treated participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 8
percentage of participants | 0 [0 to 31]

ADVERSE EVENTS:
Time Frame: Assessed on treatment continuously on treatment up to 165 days.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (N=8)
Hypothyroidism (Endocrine disorders) | 4
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 6
Pain (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Penile infection (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1
Dyspnea (Skin and subcutaneous tissue disorders) | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2
Skin/subcutaneous tissue disorders; Other (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
The study is limited by the small sample size and single-arm design along with early termination given slow accrual, lack of response and poor tolerability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No